CLINICAL TRIAL: NCT07341399
Title: Effects of EAA Consumption on Recovery and Rehabilitation in Adult Spinal Deformity (ASD) Patients Undergoing Surgery
Brief Title: Essential Amino Acid Supplementation in Adult Spinal Deformity Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 299302
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Adult Spinal Deformity
Keywords: essential amino acids; protein balance

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the effects of essential amino acid (EAA) supplementation on recovery and rehabilitation outcomes in adults undergoing corrective surgery for adult spinal deformity (ASD). Participants will be randomized to receive either an EAA supplement or an isocaloric placebo beginning two weeks prior to surgery and continuing for three months postoperatively.
  The primary objectives are to determine whether perioperative EAA supplementation improves muscle protein turnover and enhances functional recovery compared with placebo. Outcomes will include measures of muscle protein kinetics using stable isotope techniques, body composition, functional performance (handgrip strength and six-minute walk test), and clinical recovery outcomes during postoperative rehabilitation.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Essential Amino Acid Supplement Group (Experimental)
  Interventions: Dietary Supplement: Essential Amino Acid Supplement by Amino Co
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Essential Amino Acid Supplement by Amino Co — This intervention will be EAA supplementation of 15g twice a day for two weeks before surgery and then 12 weeks post-surgery in individuals diagnosed with ASD
  Arms: Essential Amino Acid Supplement Group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This will be a randomized double-blind placebo controlled clinical trial to determine if supplementing with essential amino acids (EAAs) for two weeks prior to, and 3 months after corrective spinal surgery in adults with spinal deformity can stimulate greater muscle protein turnover and whole-body protein balance, and enhance recovery after surgery when compared to a calorie matched placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, 40 to 65 years old
* Diagnosed with adult spinal deformity
* Scheduled for ASD corrective procedure at UAMS (>2 weeks prior to surgery)
* Live near Little Rock and scheduled to attend physical therapy in Little Rock
* COVID-19 negative and/ or asymptomatic

Exclusion Criteria:

* Subject who does not/will not eat animal protein sources.
* Diagnosed metabolic or hormonal disease (i.e., renal, cardiovascular, thyroid, polycystic ovary syndrome, or type I/II diabetes mellitus).
* Currently pregnant.
* Gave birth or was lactating within previous 12 months.
* History of chemotherapy or radiation therapy for cancer in the 6 months prior to enrollment.
* Clinically significant weight gain or loss (>5% change) in the last 12 months.
* Consuming metabolism-altering drugs or medications (i.e., corticosteroids, stimulants, insulin).
* Diagnosis of autoimmune disease
* Currently receiving androgen (e.g., testosterone) or anabolic (e.g., GH, IGF-I) therapy.
* Diagnosis of muscular degenerative/dystrophy disease
* Unwilling to fast overnight.
* Unwilling to avoid using other protein or amino-acid supplements during participation.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | 24 hours
  Mixed muscle protein synthesis expressed as the fractional synthetic rate.

SECONDARY OUTCOMES:
Body Composition | 12 weeks
  Body composition via DEXA will be used to examine lean body mass, fat mass, and bone mineral density. Bioelectrical impedance analysis will be used to determine total body water and muscle quality
Handgrip Strength & Walking Ability | 12 weeks
  Hand grip strength in kg and 6-min walk test ability will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Shiloah Kviatkovsky, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No